CLINICAL TRIAL: NCT00256477
Title: A Controlled Breathing Course Promoting Social and Emotional Health for Vietnam Veterans With Chronic Posttraumatic Stress Disorder - A Randomised Controlled Trial
Brief Title: A Controlled Breathing Course for Social & Emotional Health for Vietnam Veterans With Chronic PTSD-RCT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Queensland (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: SKY - PTSD; Ethics approval 2005000320
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Last update posted 2005-11-21 (Estimated); Status verified 2005-03

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

INTERVENTIONS:
Behavioral: Sudarshan KRIYA Breathing Technique

SUMMARY:
The main aim of this project is to evaluate the use of a specific Yoga technique of controlled breathing in Vietnam War Veterans with chronic posttraumatic stress disorder. This method is currently the subject of a United States grant application to formally test American War Veterans from Afghanistan and Iraq. Drs Gerbarg and Brown are collaborating with The Bay Pines Veterans Administration Medical Center in Florida to develop a study of this course for treatment of American veterans returning from Afghanistan and Iraq. Elements of this method have been used on a variety of populations. Whilst this is a multi-component intervention, it is postulated that the most active ingredient in the program is a specific Yoga breathing technique called Sudarshan Kriya (SK).

DETAILED DESCRIPTION:
The main aim of this project is to evaluate the use of a specific Yoga technique of controlled breathing in Vietnam War Veterans with chronic posttraumatic stress disorder. This method is currently the subject of a United States grant application to formally test American War Veterans from Afghanistan and Iraq. Drs Gerbarg and Brown are collaborating with The Bay Pines Veterans Administration Medical Center in Florida to develop a study of this course for treatment of American veterans returning from Afghanistan and Iraq. Elements of this method have been used on a variety of populations. Whilst this is a multi-component intervention, it is postulated that the most active ingredient in the program is a specific Yoga breathing technique called Sudarshan Kriya (SK).

This program has been developed by Sri Sri Ravi Shankar, chief yoga teacher and Head of The Art of Living Foundation (Ravishankar 2002). Further, this method has been applied widely for the treatment of Acute Stress Disorder and Posttraumatic Stress Disorder in individual cases (Gerbarg and Brown 2005Direct communication). For example, this controlled breathing program has been reported to have relieved posttraumatic stress disorder (PTSD) in large groups of people affected by mass disasters such as war (Kosovo, Bosnia, Iraq and Sudan) (Biswas 2004; Joseph 2004; Luedemann 2004), terrorism (New York City 9/11) (Anonymous 2001b), (Kashmir, India, Israel) and natural disasters (Gujurat earthquake, 2000) (Anonymous 2001a) Iran flood, Asian Tsunami. This controlled breathing program is reported to have also helped police (Slovenia, India, Washington, DC) and military personnel (Iraq) (cited in Gerbarg and Brown 2004), (Gerbarg 2005Personal communication). Pilot studies conducted by the Principal Investigator using similar techniques showed positive health results for Vietnam Veterans with PTSD in Australia (Carter and Byrne 2004). However, although randomized clinical trials have been performed for depression with good effect

ELIGIBILITY:
Inclusion Criteria:

* suffering chronic post traumatic stress disorder tested by CAPS
* Vietnam Veteran
* Adequate Cognition

Exclusion Criteria:

* Inadequate cogition
* suicidality
* psychosis
* substance abuse other than alcohol

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-03; Study Completion 2005-10

PRIMARY OUTCOMES:
Reduce the symptoms of PTSD
Reduce the comorbid conditions of Depression and alcohol dependence

CONTACTS AND LOCATIONS:
Overall Officials: Dr Janis J CARTER, MBBS FRANZCP, Principal Investigator — The University of Queensland

REFERENCES:
- See also: History of Trials thus far — http://www.therapywithyoga.com